CLINICAL TRIAL: NCT02638961
Title: Inspiratory Muscle Training and Functional Electrical Stimulation for Treatment of Heart Failure With Preserved Ejection Fraction
Brief Title: Inspiratory Muscle Training and Functional Electrical Stimulation for Treatment of HFpEF
Acronym: TRAINING-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMT-FES 01
Record Dates: First submitted 2015-12-01; First posted 2015-12-23 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: heart failure with preserved ejection fraction; physical therapy; exercise capacity; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard treatment (Placebo Comparator): Only standard medical treatment
  Interventions: Other: Standard treatment
- IMT group (Active Comparator): Standard medical treatment associated to Inspiratory muscle training
  Interventions: Other: IMT
- FES group (Active Comparator): Standard medical treatment associated to functional electrostimulation of both legs for 45 minutes a day, 2 days per week for a total of 12 weeks.
  Interventions: Other: FES
- IMT+FES group (Active Comparator): Standard medical treatment associated to combination of inspiratory muscle training and functional electrostimulation of both legs
  Interventions: Other: IMT; Other: FES

INTERVENTIONS:
Other: IMT — Patients allocated to IMT arm will receive standard medical treatment and will be instructed to train at home twice daily, for 20 minutes each session, and during 12 weeks using a threshold inspiratory muscle trainer (Threshold IMT®, Respironics Inc.). All of them will be instructed by a respiratory therapist and educated to maintain a diaphragmatic breathing during the training period. The subjects start breathing at a resistance equal to 25-30% of their maximal inspiratory pressure (MIP) for 1 week. The respiratory therapist examines the patients at weekly intervals by checking the diary card and measuring their MIP each time. The resistance is modified each session according to their 25-30% of their MIP measured.
  Other Names: Inspiratory muscular training
  Arms: IMT group; IMT+FES group
Other: FES — Patients allocated to FES arm will receive standard medical treatment and will be trained in a FES program of both legs by a physiotherapist for 45 minutes a day, 2 days per week for a total of 12 weeks. Eight adhesive electrodes are positioned on the skin over the quadriceps and gastrocnemius muscles of both legs. The stimulator is configured to deliver a direct electrical current at 25 Hz for 5 seconds followed by a 5-second rest. The intensity of the stimulation is adjusted to achieve a visible muscle contraction without discomfort.
  Other Names: Functional electrostimulation of lower limbs
  Arms: FES group; IMT+FES group
Other: Standard treatment — Patients allocated to this arm will not receive any physical therapy, only standard medical treatment. They will be checked weekly by a physiotherapist who measures their maximal inspiratory mouth pressure each time.
  Arms: Standard treatment

SUMMARY:
Heart failure (HF) with preserved ejection fraction (HFpEF) has become the most prevalent form of HF in developed countries. Despite its increasing in prevalence, there is no evidence-based effective therapy for HFpEF The purpose of this study was to evaluate whether inspiratory muscle training (IMT), functional electrical stimulation (FES), or combination of both improve exercise capacity as well as left ventricular diastolic function, biomarkers' profile, quality of life (QoL) and prognosis in patients with HFpEF.

DETAILED DESCRIPTION:
This study was designed as a prospective, controlled, randomized, four-armed, efficacy trial of patients with the diagnosis of HFpEF and New York Heart Association functional class II-III/IV, diagnosed according to criteria of the European Society of Cardiology. A computer-generated randomization scheme was used to allocate participants (in a 1:1:1:1 ratio) to receive: 1) a home-based 12-week program of inspiratory muscle training (IMT) or; 2) a 12-week program of functional electrical stimulation (FES) of lower limb muscles or; 3) standard treatment (ST) alone or; 4) combination of IMT and FES. The study is being conducted in a single center in Spain. Independently of staggered entry, the minimum duration of a patient's participation is 6 months (from first to last visit). All patients will provide signed informed consent and the protocol has been approved by the research ethics committee of our center in accordance with the principles of the Declaration of Helsinki and national regulations.

Study population Candidate patients are selected from the outpatient's clinics of HF of the Hospital Clínico Universitario of Valencia.

Study objectives The primary endpoint of the study is a clinical endpoint of three and six months change in peak oxygen uptake (peak VO2).

Secondary endpoints are three and six month changes in echocardiogram parameters, QoL and prognostic biomarkers. The investigators also will specifically focus on number of episodes of worsening HF at 6 months:

1. Change in E/e' after three and six months.
2. Change in left atrial volume index after three and six months.
3. Change in health-related QoL measured by the Minnesota Living With Heart Failure Questionnaire (MLHF) after three and six months.
4. Change in natriuretic peptide (NT-proBNP) after three and six months.
5. Change in minute ventilation/carbon dioxide production (VE/VCO2) slope after three and six months.
6. Number of episodes of acute HF hospitalizations and number of episodes of worsening HF not requiring hospitalization at 6 months.

Intervention

Eligibility assessment and screening visit After reviewing the inclusion/exclusion criteria and signing the informed consent form, a comprehensive medical history, physical examination, anthropometry and examination tests will be performed. The examination tests include: electrocardiogram (ECG) echocardiography, cardiopulmonary exercise testing (CPET), 6-minute walk test (6-MWT), inspiratory muscle function test, QoL assessment by the Minnesota Living With Heart Failure Questionnaire (MLHF) and blood samples for a panel of baseline biomarkers.

Finally, patients are randomized (1:1:1:1) to four groups: 1) ST alone or; 2) a home-based 12-week program of IMT or; 3) a 12-week program of FES or; 4) combination of IMT and FES (IMT+FES) during 12 weeks.

12-week and six months visits All patients will be evaluated after 12-week supervised training, and six months after randomization. Evaluation will include medical history, physical examination, anthropometry and functional and QoL assessment tests (ECG, CPET, 6-MWT, inspiratory muscle function test, MLHF and blood tests).

ELIGIBILITY:
Inclusion Criteria:

* Previous history of symptomatic heart failure NYHA (New York Heart Association )functional class ≥II with Normal left ventricular ejection fraction:

  * ejection fraction >0.50 by Simpson method
  * end-diastolic diameter <60 mm
* Structural heart disease:

  * left ventricle hypertrophy/left atrial enlargement and/or
  * diastolic dysfunction estimated by 2D echocardiography
* Previous admission for acute heart failure
* Clinical stability, without hospital admissions in the past 3 month

Exclusion Criteria:

* Perform a valid baseline exercise test
* Significant primary moderate to severe valvular disease
* Acute coronary syndrome or cardiac surgery within the previous three months
* Signs of ischemia during cardiopulmonary exercise testing
* Significant primary pulmonary disease; including pulmonary arterial hypertension, chronic thromboembolic pulmonary disease or chronic obstructive pulmonary disease
* Any other comorbidity with an expectancy of life less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Functional capacity measured as peak oxygen uptake (peak VO2) in ml/min/kg . | changes at 12 weeks and 6 months
  Maximal functional capacity will be evaluated with an incremental and symptom-limited cardiopulmonary exercise testing (CORTEX Metamax 3B) on a bicycle ergometer, beginning with a workload of 10 W and increasing stepwise at 10-W increments every 1 min. During exercise, patients were continuously monitored with twelve-lead electrocardiogram and blood pressure measurements every 2 min. Gas exchange data and cardiopulmonary variables were averaged every 10 seconds values. Peak VO2 is considered the highest value of VO2 during the last 20 s of exercise.
  The improvement > of 10% in peak VO2 will be considered clinically meaningful

SECONDARY OUTCOMES:
Functional capacity measured as distance walked in 6 minutes | changes at 12 weeks and 6 months
  Patients will be instructed to cover the maximum distance (meters) possible in six minutes, at a self-graded walking speed, pausing to rest when needed. Each subject will undergo 4 tests. The goal of the first one was to allow the patient to familiarize with the test.
Change in echocardiographic parameter of diastolic disfunction: e' septal (cm/s) | changes in rest at 12 weeks and 6 months
  Doppler echocardiogram examination of e' septal (cm/s) will be performed under resting conditions using 2D echocardiography (iE33, Philips). e' septal (cm/s) parameter will be measured according to current guidelines of the European Society of Echocardiography:
  Only significant improvements in this parameter will be considered
Change in echocardiographic parameter of diastolic disfunction: left atrial volume index (mm/m2) | changes in rest at 12 weeks and 6 months
  Doppler echocardiogram examination of left atrial volume index (mm/m2) will be performed under resting conditions using 2D echocardiography (iE33, Philips). Left atrial volume index (mm/m2) will be measured according to current guidelines of the European Society of Echocardiography.
  Only significant improvements in this parameter will be considered
Change in echocardiographic parameter of diastolic disfunction: E/e' ratio | changes in rest at 12 weeks and 6 months
  Doppler echocardiogram examination of E/e' ratio will be performed under resting conditions using 2D echocardiography (iE33, Philips). E/e' ratio parameter will be measured according to current guidelines of the European Society of Echocardiography.
  Only significant improvement in this parameter will be considered
Change in health-related QoL | changes at 12 weeks and 6 months
  Change in health-related QoL will be measured by the Minnesota Living With Heart Failure Questionnaire (no units) Only significant improvements in these parameters will be considered
Number of rehospitalizations or worsening HF at 6 months | changes at 6 months
  Number of episodes of acute HF hospitalizations and number of episodes of worsening HF not requiring hospitalization at 6 months among different arms.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Palau, M.D., PhD, Principal Investigator — Universitat Jaume I; Eloy Domínguez, M.D, Study Director — Universitat Jaume I; Julio Núñez, M.D., PhD, Study Chair — Universitat de Valencia
Locations (1):
- Hospital clínico universitario de Valencia, Valencia, Spain

REFERENCES:
- [Background] Palau P, Dominguez E, Nunez E, Schmid JP, Vergara P, Ramon JM, Mascarell B, Sanchis J, Chorro FJ, Nunez J. Effects of inspiratory muscle training in patients with heart failure with preserved ejection fraction. Eur J Prev Cardiol. 2014 Dec;21(12):1465-73. doi: 10.1177/2047487313498832. Epub 2013 Jul 17. PMID 23864363
- [Background] Palau P, Nunez E, Dominguez E, Sanchis J, Nunez J. Physical therapy in heart failure with preserved ejection fraction: A systematic review. Eur J Prev Cardiol. 2016 Jan;23(1):4-13. doi: 10.1177/2047487314562740. Epub 2014 Dec 8. PMID 25488549
- [Derived] Palau P, Dominguez E, Lopez L, Ramon JM, Heredia R, Gonzalez J, Santas E, Bodi V, Minana G, Valero E, Mollar A, Bertomeu Gonzalez V, Chorro FJ, Sanchis J, Lupon J, Bayes-Genis A, Nunez J. Inspiratory Muscle Training and Functional Electrical Stimulation for Treatment of Heart Failure With Preserved Ejection Fraction: The TRAINING-HF Trial. Rev Esp Cardiol (Engl Ed). 2019 Apr;72(4):288-297. doi: 10.1016/j.rec.2018.01.010. Epub 2018 Mar 16. English, Spanish. PMID 29551699